CLINICAL TRIAL: NCT04170257
Title: Performance of White Light, Narrow Band Imaging and Iodine Staining Endoscopy in the Diagnosis of Esophageal Squamous Epithelium Lesions: A Multicenter Clinical Study in China
Brief Title: Performance of White Light, NBI and Iodine Staining Endoscopy in the Diagnosis of Esophageal Lesions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Yang Ke, Professor, Peking University Cancer Hospital & Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2018KT111
Record Dates: First submitted 2019-11-17; First posted 2019-11-20 (Actual); Last update posted 2019-11-20 (Actual); Status verified 2019-11

CONDITIONS: Mild Dysplasia of Esophagus; Moderate Dysplasia of Esophagus; Severe Dysplasia of Esophagus; Carcinoma in Situ of Esophagus; Esophageal Squamous Cell Carcinoma
Keywords: Esophageal Squamous Cell Carcinoma; Population-level screening; Narrow Band Imaging; Iodine Staining; Sensitivity and Specificity
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma; Hypersensitivity | interventions — Narrow Band Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Opportunistic screening cohort (Experimental): This opportunistic screening cohort is constructed among patients aged 45-69 years who undergo endoscopic examinations at the endoscopy center in any of the five hospitals included in this study. Enrolled participants are requested to complete a computer aided one-on-one questionnaire regarding demographic factors, smoking and alcohol drinking status, dietary habits，digestive tract symptoms and family history of ESCC. Then experienced endoscopists will perform the upper gastrointestinal endoscopic examination for each participant, and the entire esophagus will be visually examined with the white light, NBI and iodine staining endoscopic examination.
  Interventions: Diagnostic Test: Endoscopic examination using white light, NBI and iodine staining

INTERVENTIONS:
Diagnostic Test: Endoscopic examination using white light, NBI and iodine staining — Participants' esophagus will be examined by three commonly used diagnostic techniques in the order of : 1. White light endoscopy (WLE); 2. Narrow Band Imaging (NBI) and 3. Iodine Staining Endoscopy (ISE) with 1.2% Lugol's iodine solution. The required observation time is no less than 1 minute for WLE and 2 minutes for NBI and ISE. Endoscopic images of each participant are routinely captured at every 5 centimeters in the esophagus, and information is recorded in detail for each focal lesion. Biopsies are taken from all visually abnormal areas found by any one of the three techniques, histopathologic diagnoses are rendered by two pathologists according to standard criteria and discrepancies are adjudicated by consultation. The recorded endoscopic images for each biopsied lesion are read by two trained researchers and the visualized feature of lesions are decomposed into several indicators (e.g. size, shape, color, and border of lesions) .

SUMMARY:
The investigators aim to evaluate the performance of Narrow Band Imaging (NBI) endoscopy in Esophageal Squamous Cell Carcinoma (ESCC) screening, as compared to the currently used White Light Endoscopy (WLE) and Lugol's Iodine Staining Endoscopy (ISE). NBI is a simple, safe and non-invasive technique, which can provide real-time optical staining for suspicious lesions. This trial is designated to enroll 10000 participants from five centers located in different regions (North, West and South) in China, which would provide real-world evidence for the recommendation of endoscopic diagnostic technique used in ESCC screening projects.

ELIGIBILITY:
Inclusion Criteria:

* Patients seek for endoscopic examinations at the endoscopy center in any of the five hospitals included in this study
* Aged 45-69 years
* Have entire esophagus
* Provide written informed consent and leave personal identification and contact information

Exclusion Criteria:

* Have contraindications to endoscopic examination (Including but not limited to severe arrhythmia, myocardial infarction, heart failure, hemiplegia, asthma, severe hypertension (≥ 180 / 110mmHg), psychosis, etc )
* Have a history of drug allergy
* Have a history of upper gastrointestinal surgery
* Have a history of radiotherapy or chemotherapy

Ages: 45 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10000 (Estimated)
Dates: Start 2019-10-18 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of WLE, NBI and ISE in the diagnosis of mild, moderate, severe dysplasia and above lesions in esophagus | 0 days
  Sensitivity of WLE, NBI and ISE, taking results from histopathological analysis of the biopsy specimens as the golden standard.
Specificity of WLE, NBI and ISE in the diagnosis of mild, moderate, severe dysplasia and above lesions in esophagus | 0 days
  Specificity of WLE, NBI and ISE, taking results from histopathological analysis of the biopsy specimens as the golden standard.
Positive predictive value (PPV) of WLE, NBI and ISE in the diagnosis of mild, moderate, severe dysplasia and above lesions in esophagus | 0 days
  PPV of WLE, NBI and ISE, taking results from histopathological analysis of the biopsy specimens as the golden standard.
Negative predictive value (NPV) of WLE, NBI and ISE in the diagnosis of mild, moderate, severe dysplasia and above lesions in esophagus | 0 days
  NPV of WLE, NBI and ISE, taking results from histopathological analysis of the biopsy specimens as the golden standard.

SECONDARY OUTCOMES:
Weight of each visualized abnormal feature of lesions | 0 days
  The estimated odds ratio of each decomposed graphic abnormal features of lesions, taking "severe dysplasia and above" diagnosed via histopathological analysis as the outcome events.
Discrimination of visualized abnormal features | 0 days
  The area under the curve (AUC) of visualized graphic abnormal features for predicting severe dysplasia and above lesions.

CONTACTS AND LOCATIONS:
Overall Officials: Mengfei Liu, PhD, Study Director — Peking University Cancer Hospital & Institute
Locations (5):
- China (5):
  - Beijing Friendship Hospital, Beijing, Beijing Municipality
  - Shantou University Medical College Affiliated Cancer Hospital, Shantou, Guangdong
  - Anyang Cancer Hospital, Anyang, Henan
  - People's Hospital of Hua County, Henan Province, Anyang, Henan
  - People's Hospital of Ningxia Hui Autonomous Region, Yinchuan, Ningxia